CLINICAL TRIAL: NCT01960946
Title: Galectin-3 Inhibition With Modified Citrus Pectin in Hypertension
Brief Title: Galectin-3 Blockade in Patients With High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jennifer En-Sian Ho M.D., Assistant in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015P0023402; K23HL116780 (NIH)
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
Keywords: Hypertension; Galectin 3; Fibrosis; Vascular Stiffness; Echocardiography
MeSH Terms: conditions — Hypertension; Fibrosis | interventions — citrus pectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified Citrus Pectin (MCP) (Active Comparator): Dietary Supplement: Modified Citrus Pectin (MCP, PectaSol-C), 5 grams by mouth three times a day
  Interventions: Dietary Supplement: Modified Citrus Pectin (MCP) vs placebo
- Placebo (Placebo Comparator): Matched placebo 5 grams by mouth three times a day
  Interventions: Dietary Supplement: Modified Citrus Pectin (MCP) vs placebo

INTERVENTIONS:
Dietary Supplement: Modified Citrus Pectin (MCP) vs placebo — 5 grams by mouth three times a day
  Other Names: MCP; PectaSol-C

SUMMARY:
This study will investigate if Modified Citrus Pectin (MCP) can help people with high blood pressure. MCP is a dietary supplement that is derived from plants, and therefore is not subject to approval by the U.S. Food and Drug Administration (FDA). However, MCP has been deemed as 'generally regarded as safe' by the FDA.

This study will examine whether Modified Citrus Pectin (MCP) can help people with high blood pressure. The study will help understand how MCP may affect the risk for heart disease in patients with high blood pressure.

DETAILED DESCRIPTION:
Gal-3 appears to be a potential mediator of cardiac fibrosis, preceding the development of clinical heart failure. In this study, we seek to identify individuals at risk for the development of heart failure based on clinical hypertension and elevated Gal-3 concentrations. Participants will be randomized to receive a Gal-3 inhibitor (MCP) or placebo. The primary outcome will be the effect on collagen metabolism, and secondary outcomes include echocardiographic measures of cardiac structure and function, and non-invasive measures of vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-70 years
* Physician diagnosed hypertension on stable therapy for 3 months
* Elevated galectin-3 level (above sex-specific median based on Framingham Heart Study measures)
* Able to understand the protocol and provide informed consent in English

Exclusion Criteria:

* Uncontrolled hypertension, defined as systolic blood pressure > 170mmHg, diastolic blood pressure > 100mmHg
* Evidence of secondary hypertension
* History of heart failure, coronary artery disease, stroke, atrial fibrillation
* Left ventricular ejection fraction < 45% on echocardiography
* Use of aldosterone antagonists
* History of liver cirrhosis
* History of pulmonary fibrosis
* Kidney dysfunction, defined as estimated glomerular filtration rate < 45 ml/min/1.73m2
* Anemia, defined as hematocrit < 37% in men and < 34% in women
* Use of chelating agents
* History of Active cancer or malignancy
* Known pregnancy, those unwilling to avoid pregnancy during the course of the study, or women currently breastfeeding
* Hyperkalemia on screening labs, defined as potassium >5.2
* Anticipated inability to complete or comply with study protocol
* History of angioedema

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-10; Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change in markers of collagen metabolism | Baseline and 6 months
  Primary aim will be change in markers of collagen metabolism (PICP, PIIICP, ICTP, TIMP-1) in MCP versus placebo groups over 6 months of treatment.

SECONDARY OUTCOMES:
Change in galectin-3 level | Baseline and 6 months
  Changes in galectin-3 level from baseline until 6 months will be compared between MCP and placebo groups
Changes in cardiac structure and function | Baseline and 6 months
  Changes in cardiac structure and function will be examined using 2-D echocardiography and tissue Doppler imaging. This will include changes in left ventricular mass, dimensions, left atrial size, and left ventricular diastolic function.
Changes in arterial stiffness | Baseline and 6 months
  We will examine changes in arterial stiffness (including augmentation index, carotid-femoral pulse-wave velocity) from baseline to 6 months in the MCP and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Ho, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lau ES, Liu E, Paniagua SM, Sarma AA, Zampierollo G, Lopez B, Diez J, Wang TJ, Ho JE. Galectin-3 Inhibition With Modified Citrus Pectin in Hypertension. JACC Basic Transl Sci. 2021 Jan 6;6(1):12-21. doi: 10.1016/j.jacbts.2020.10.006. eCollection 2021 Jan. PMID 33532663